CLINICAL TRIAL: NCT04106973
Title: Identification of Biomarkers for the Early Detection of Mesothelioma
Brief Title: Mesothelioma Early Detection by VOCs
Acronym: MED-VOC
Status: Terminated | Type: Observational
Why Stopped: Recruitment suspended secondary to social distancing directive associated with Covid-19
Sponsor: Henry Ford Health System (Other)
Collaborators: International Association of Heat and Frost Insulators and Allied Workers (Other); Owlstone Ltd (Industry); Fujirebio Diagnostics, Inc. (Industry)
Responsible Party: Principal Investigator, David Svinarich, Ph.D., VP-Research, Henry Ford Health System
Other Study IDs: 1432436
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Pleural Mesothelioma; Asbestos Exposure; Pleural Plaque
Keywords: Pleural Mesothelioma; Bilateral Pleural Plaques; Asbestos Exposure; Exhaled breath analysis; VOCs
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Exhaled breath collected in four stainless steel sorbent tubes and serum specimen and serum specimen from each subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pleural mesothelioma: Participants with all types of histologically identified pleural mesothelioma prior to, subsequent to,or concurrent with treatment.
- Asbestos exposed without pleural mesothelioma: Participants with asbestos exposure radiographically confirmed by the presence of bilateral pleural plaques or bilateral pleural thickening and without presence of pleural mesothelioma.

SUMMARY:
This is a two phase study, The first phase (phase 1) will identify potential biomarkers among asbestos exposed individuals with pleural mesothelioma. The second phase (phase 2), is a double blinded case-matched controlled study to determine the predictive capability, sensitivity, and specificity of these biomarkers in detecting early stage pleural mesothelioma. Biomarkers in the form of volatile organic compounds (VOC) in exhaled breath samples from subjects with either pleural mesothelioma or pleural plaques, will be evaluated. A biomarker present in serum will also be concurrently evaluated in the same cohort. The soluble serum biomarker mesothelin related peptides (SMRP), which has been posited as a biomarker for mesothelioma, will be analyzed for its relationship to the breath VOC profile.

DETAILED DESCRIPTION:
Mesothelioma is a rare, aggressive and treatment-resistant disease and, in the United States, is caused almost exclusively by exposure to asbestos fibers. There is often a lengthy latency period of 40-50 years between exposure and disease onset. The median age of diagnosis is 65 years while the median survival time after diagnosis of pleural mesothelioma without treatment is 9 months. Symptoms, where present, may be non-specific, which further contributes to delayed diagnosis.

In this study, the volatile organic compound (VOC) profile of exhaled breath from subjects with histologically confirmed mesothelioma will be compared against case-matched control subjects with bilateral pleural plaques or bilateral pleural thickening. Putative markers will then be tested against a blinded cohort to test predictive value of the markers.

This study seeks to identify markers for mesothelioma using a non-invasive technique which samples volatile organic compounds (VOC) in the breath of test subjects (Owlstone Medical Ltd, Cambridge, England).

A comparison of the participant's VOC profile will be made with an FDA-approved, serum-based assay (Lumipulse Mesomark®, Fujirebio Diagnostics Inc., Malvern, PA) of the participant's soluble mesothelin related peptides (SMRP) to discern parameters of efficacy..

ELIGIBILITY:
Inclusion Criteria

* Male or Female over 18 years of age
* Clinical diagnosis of pleural mesothelioma or presence of pleural plaques on X-Ray
* Documented exposure to asbestos
* Must be able to provide breath sample
* Must be able to provide relevant medical information

Exclusion Criteria

* Presence of malignancies other that mesothelioma within the past 6 months
* Treatment for any malignancies other than mesothelioma within the past 6 months
* Inability to provide past clinical information
* Inability to perform breath collection procedure
* Smoking or consuming alcohol within two hours of conducting breath collection procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with histologically confirmed pleural mesothelioma, and individuals with an asbestos exposure and radiological evidence of bilateral pleural plaques or pleural thickening without evidence of mesothelioma. The majority of asbestos exposed participants with bilateral pleural thickening or pleural plaques and no mesothelioma will be active or retired members of the International Association of Heat and Frost Insulators and Allied Workers Union.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
VOC markers in breath samples. Predictive capability, sensitivity and specificity of biomarkers present in volatile organic compounds (VOC) for the early detection of pleural Mesothelioma in patients exposed to asbestos. | At study completion, approximately 2 years
  Predictive capability, sensitivity and specificity of biomarkers present in volatile organic compounds (VOC) for the early detection of pleural Mesothelioma in patients exposed to asbestos.

SECONDARY OUTCOMES:
Predictive capability, sensitivity and specificity of Soluble Mesothelin Related Peptides (SMRP) in serum when combined with VOC biomarkers for pleural mesothelioma. | At study completion, approximately 2 years
  Determine the additive predictive capability, sensitivity and specificity of SMRP serum biomarkers with VOC biomarkers for the early detection of pleural mesothelioma

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Harbut, MD, MPH, Principal Investigator — Ascension Providence Hospital, Southfield; David M Svinarich, PhD, Principal Investigator — Ascension Providence South East Michigan
Locations (1):
- Consultants in Sleep and Pulmonary Medicine, Farmington Hills, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Gennaro G, Dragonieri S, Longobardi F, Musti M, Stallone G, Trizio L, Tutino M. Chemical characterization of exhaled breath to differentiate between patients with malignant plueral mesothelioma from subjects with similar professional asbestos exposure. Anal Bioanal Chem. 2010 Dec;398(7-8):3043-50. doi: 10.1007/s00216-010-4238-y. Epub 2010 Oct 6. PMID 20924566
- [Background] Oliver LC, Welch LS, Harbut MR. Comparison of B readers' interpretations of chest radiographs for asbestos related changes. Acad Radiol. 2004 Dec;11(12):1397-9; author reply 1402-4. doi: 10.1016/j.acra.2004.09.010. No abstract available. PMID 15596380

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT04106973/Prot_SAP_000.pdf